CLINICAL TRIAL: NCT01280383
Title: Non-invasive Neurally Adjusted Ventilatory Assist (niNAVA) After Extubation: Proposal for a Crossover-randomized Feasibility Trial
Brief Title: Non-invasive Neurally Adjusted Ventilatory Assist
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study does not meet the new legal requirements set forth in the Human Research Act
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BE KEK 123/10
Record Dates: First submitted 2011-01-10; First posted 2011-01-20 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Failure
Keywords: non-invasive ventilation; diaphragm; electrical activity; neurally adjusted ventilatory assist; critically ill patients
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Interactive Ventilatory Support; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- non-invasive NAVA (Experimental): application of non-invasive NAVA in critically ill patients
  Interventions: Device: non-invasive neurally adjusted ventilatory assist

INTERVENTIONS:
Device: non-invasive neurally adjusted ventilatory assist — non-invasive neurally adjusted ventilatory assist in critically ill patients
  Other Names: neurally adjusted ventilatory assist; non-invasive ventilation

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a new concept of mechanical ventilation. NAVA delivers assistance to spontaneous breathing based on the detection of the electrical activity of the diaphragm. The investigators will study the effects of non-invasive NAVA on respiratory muscle unloading critically ill patients.

DETAILED DESCRIPTION:
To assess the effects of non-invasive NAVA on respiratory muscle unloading in critically ill patients

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years
* History of chronic obstructive lung disease
* Invasive mechanical ventilation for more than 12 hours
* Planned extubation according to the weaning protocol of our clinic
* Informed consent obtained from a next of kin
* Enrollment approval from a neutral physician neither participating in the study nor in the clinical treatment of the patient

Exclusion Criteria:

* Tracheostomy
* Facial or cranial trauma or surgery
* Oral, esophageal, diaphragmatic or gastric trauma or surgery
* Contraindication to insertion of a nasogastric tube (e. g. malformation, esophageal varices, esophageal perforation or rupture, Zenkers diverticulum, severe bleeding disorder)
* Uncooperative state and combativeness not responding to low levels of sedatives
* Neurological disease possibly influencing the brainstem respiratory centre, such as but not limited to: intracerebral, subarachnoidal or subdural hemorrhage, cerebral infarction, possible hypoxic encephalopathy
* Next of kin refuses informed consent
* Pregnancy. In female patients between 18 and 60 years of age, a pregnancy test will be performed.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
patient-ventilator synchrony | outcomes are assessed at the end of each experimental period, i.e. every 20-30 minutes

SECONDARY OUTCOMES:
changes in respiratory pattern | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Brander, MD, Principal Investigator — University Hospital (Inselspital) and University of Bern

REFERENCES:
- [Background] Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med. 1999 Dec;5(12):1433-6. doi: 10.1038/71012. No abstract available. PMID 10581089